CLINICAL TRIAL: NCT00288951
Title: Phase III Safety and Efficacy Study to Evaluate a Glaucoma Therapy in Open-Angle Glaucoma or Ocular Hypertension Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-04-17
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2009-09

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost

INTERVENTIONS:
Drug: Travoprost 0.004% with and without BAK

SUMMARY:
The purpose of this study is to determine the safety and IOP-lowering ability of a glaucoma therapy in patients with open-angle glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects of either sex and any race 18 years or older with open-angle glaucoma or ocular hypertension. Patients with logMAR visual acuity not worse than 0.6 in either eye or any clinically relevant ophthalmic/systemic condition will be excluded.

Exclusion Criteria:

* See Inclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Actual)
Dates: Start 2004-10; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)